CLINICAL TRIAL: NCT04012814
Title: Clinical Evaluation of the Safety and Efficacy of a 1060 nm Diode Laser, Pulsed ElectroMagnetic Fields and Vacuum Assisted Multipolar Radio Frequency for Non-invasive Fat Reduction of the Abdomen and Flanks
Brief Title: Clinical Evaluation of a 1060 nm Diode Laser, PEMF and Vacuum Assisted MP RF for Non-invasive Fat Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL0319
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Adipose Tissue Atrophy
Keywords: fat; abdomen fat; flank fat; body contouring
MeSH Terms: conditions — Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Intervention Model Description: Up to 200 subjects will be enrolled in the study to receive 3 Diode and 3 RF treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Subject treatment group (Experimental): Treatment group receiving 3 diode treatments and 3 RF/PEMF treatments at Week 0, 8 and 16 with a follow-up at Week 24.
  Interventions: Device: Venus Bliss

INTERVENTIONS:
Device: Venus Bliss — The FDA cleared device (Venus Bliss™) is a non-invasive medical aesthetic device designed for body contouring. The device is comprised of a console, four 1060 nm diode laser applicators (60 mm x 60 mm). A belt is included to allow the operator to secure the laser applicators on the lipolysis treatment area, allowing hands free operation. The device uses vacuum assisted radiofrequency (RF) and PEMF (pulsed electromagnetic field) technology which has been shown in clinical studies to be safe and effective in body circumferential reduction and skin tightening.

SUMMARY:
Open-label, baseline-controlled, multi-center study evaluating a 1060 nm diode laser, pulsed electromagnetic fields and vacuum assisted radio frequency for non-invasive fat reduction of the abdomen and flanks.

DETAILED DESCRIPTION:
Open-label, baseline-controlled, multi-center study evaluating a 1060 nm diode laser, pulsed electromagnetic fields, and vacuum-assisted radio frequency for non-invasive fat reduction of the abdomen and flanks. The study will enroll up to 200 subjects requesting non-invasive lipolysis of the abdomen and flanks. Each subject will receive 3 study treatments of the diode laser and 3 treatments of the pulsed electromagnetic fields and vacuum assisted radio frequency. Subjects will be followed at twelve weeks post-final diode treatment. The twelve-week post-treatment outcome will be compared to the baseline.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to read, understand and voluntarily provide written informed consent. 2. Healthy male or female, ≥ 18 years of age seeking treatment for unwanted fat in the flanks.

  3. BMI score is less than 35. 4. Agree to not making any major changes in their diet or lifestyle during the course of the study.

  5. Able and willing to comply with the treatment/follow-up schedule and requirements.

  6. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study, and have a negative Urine Pregnancy test at baseline.

Exclusion Criteria:

* 1. Pregnant in the last 3 months, intending to become pregnant, postpartum or nursing in the last 6 months.

  2. Any previous liposuction/lipo-sculpture or any type of surgical procedure in the treatment area in the past 12 months.

  3. History of immunosuppression/immune deficiency disorders (including AIDS and HIV infection) or use of immunosuppressive medications, 6 months prior to and during the course of the study.

  4. History of hyperlipidemia, diabetes mellitus, hepatitis, blood coagulopathy or excessive bleeding.

  5. Use of antiplatelet medications (81 mg acetylsalicylic acid daily permitted), anticoagulants, thrombolytics or anti-inflammatory medications within 2 weeks of treatment.

  6. Having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions.

  7. Having a permanent implant in the treatment area such as metal plates or an injected chemical substance such as silicone or parenteral gold therapy (gold sodium thiomalate).

  8. Use of medications, herbs, food supplements, and vitamins known to induce photosensitivity to light exposure at the wavelength used or history of photosensitivity disorder.

  9. Suffering from significant skin conditions in the treatment area or inflammatory skin conditions including but not limited to open lacerations, abrasions, herpes sores, cold sores, active infections.

  10. Tattoos in the treatment area. 11. Poor skin quality (severe laxity). 12. Abdominal wall, muscular abnormality or hernia on physical examination. 13. Use of retinoids such as oral isotretinoin (Accutane™) within the past six months or during course of the study.

  14. History of keloid or hypertrophic scar formation or poor wound healing in the treatment area.

  15. As per the investigator's discretion, any physical or mental condition which may make it unsafe for the subject to participate.

  16. Unable or unlikely to refrain from sun exposure, artificial tanning, including the use of tanning booths, prior to (six weeks) and during the course of the evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoni Iger, PhD, Study Director — Venus Concept LTD
Locations (5):
- United States (5):
  - Berman Skin Institute, Los Altos, California
  - Laser & Skin Surgery Medical Group, Inc, Sacramento, California
  - Batra Dermatology, Santa Monica, California
  - aFresh Medispa, Chicago, Illinois
  - UT Southwestern Medical Center Department of Plastic Surgery, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
No plan to share data with other researchers

RESULTS

PARTICIPANT FLOW:
Groups:
- Subject Treatment Group: Treatment group received 3 diode treatments and 3 RF/PEMF treatments at Week 0, 8 and 16.
  Venus Bliss: The FDA-cleared device (Venus Bliss™) is a non-invasive medical aesthetic device designed for body contouring. The device is comprised of a console, and four 1060 nm diode laser applicators (60 mm x 60 mm). A belt is included to allow the operator to secure the laser applicators on the lipolysis treatment area, allowing hands-free operation. The device uses vacuum-assisted radiofrequency (RF) and PEMF (pulsed electromagnetic field) technology which has been shown in clinical studies to be safe and effective in body circumferential reduction and skin tightening.
Period: Overall Study
Arm/Group | Subject Treatment Group
Started | 39
Completed | 31
Not Completed | 8
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Subject Treatment Group: Treatment group received 3 diode treatments and 3 RF/PEMF treatments.
  Venus Bliss: The FDA-cleared device (Venus Bliss™) is a non-invasive medical aesthetic device designed for body contouring. The device is comprised of a console, and four 1060 nm diode laser applicators (60 mm x 60 mm). A belt is included to allow the operator to secure the laser applicators on the lipolysis treatment area, allowing hands-free operation. The device uses vacuum-assisted radiofrequency (RF) and PEMF (pulsed electromagnetic field) technology which has been shown in clinical studies to be safe and effective in body circumferential reduction and skin tightening.
Arm/Group | Subject Treatment Group
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 37
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Aesthetic Appearance From Baseline
Description: Photographic evaluation by an independent, blinded reviewer with correct identification of pre-treatment baseline images when compared to post-treatment images taken at Week 24 using the Global Aesthetic Improvement Scale (GAIS). A score of 0 is no change, 1 - slight change, 2 - moderate change, 3 - dramatic change. An incorrect identification would result in a negative score (-1 for slight, -2 for moderate and -3 for dramatic change)
Time Frame: Week 24
Population: All subjects who had both Week 0 (baseline) and Week 24 (follow-up) photos.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Subject Treatment Group
Number analyzed (Participants) | 31
score on a scale | 0.97 (0.08)

2. Secondary Outcome: Subject Satisfaction: 5-Point Likert Subject Satisfaction Scale
Description: To assess subject satisfaction with treatment at the Week 24 visit using the 5-point Likert Subject Satisfaction Scale: 0 - very dissatisfied, 1 - dissatisfied, 2 - neutral, 3 - satisfied, 4 - very satisfied.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Subject Treatment Group
Number analyzed (Participants) | 31
Participants
  Very Satisfied (4) | 10
  Satisfied (3) | 11
  Neutral | 9
  Dissatisfied | 1
  Very Dissatisfied | 0

3. Secondary Outcome: Change in Fat Thickness
Description: Fat thickness was measured using ultrasound at one clinical site (14 subjects in total). Change between Week 0 and Week 24 measurements is shown.
Time Frame: Week 24
Measure: Mean (Standard Error); unit: percentage of baseline
Arm/Group | Subject Treatment Group
Number analyzed (Participants) | 14
percentage of baseline | -6.9 (1.1)

ADVERSE EVENTS:
Time Frame: Up to the 24 week follow-up visit
Groups:
- Subject Treatment Group: Treatment group received up to 3 diode treatments and up to 3 RF/PEMF treatments at Week 0, 8 and 16.
  Venus Bliss: The FDA-cleared device (Venus Bliss™) is a non-invasive medical aesthetic device designed for body contouring. The device is comprised of a console, and four 1060 nm diode laser applicators (60 mm x 60 mm). A belt is included to allow the operator to secure the laser applicators on the lipolysis treatment area, allowing hands-free operation. The device uses vacuum-assisted radiofrequency (RF) and PEMF (pulsed electromagnetic field) technology which has been shown in clinical studies to be safe and effective in body circumferential reduction and skin tightening.
Arm/Group | Subject Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 8/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subject Treatment Group (N=39)
Bruise (Skin and subcutaneous tissue disorders) | 1 (1)
Temporary Nodule (Skin and subcutaneous tissue disorders) | 6 (6)
Tenderness (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT04012814/Prot_SAP_000.pdf